CLINICAL TRIAL: NCT03998904
Title: Muscle Preservation Hamstring Graft for ACL Reconstruction: Randomized Controlled Trial
Brief Title: Muscle Preservation Hamstring Graft for ACL Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanyang University Seoul Hospital (Other)
Responsible Party: Principal Investigator, JIN KYU LEE, professor, Hanyang University Seoul Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: muscle preservation study
Record Dates: First submitted 2019-06-25; First posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Graft Healing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle preservation (Experimental): Muscle preservation for hamsting graft
  Interventions: Procedure: Muscle preservation
- None preservation (Active Comparator): No muscle preservation for hamstring graft
  Interventions: Procedure: No muscle preservation

INTERVENTIONS:
Procedure: Muscle preservation — Muscle preservation during graft preparation of hamstring graft
  Arms: Muscle preservation
Procedure: No muscle preservation — No muscle preservation during graft preparation of hamstring graft
  Arms: None preservation

SUMMARY:
* Muscle derived stem cell is a better source of stem cells than a tendon tissue
* Preservation of muscle derived stem cell may enhance bone-tendon integration and ligamentization of ACL hamstring graft

ELIGIBILITY:
Inclusion Criteria:

* Primary ACL reconstruction using autogenous hamstring graft

Exclusion Criteria:

* Combined meniscal or ligament surgery
* Combined osteoarthritis (KL grade II or more)
* chondral injury more than grade 2
* Refuse to undergo MRI

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
SNQ value of MRI | 6 months
  signal of ACL graft-signal of quadriceps tendon/singal of background

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang University Seoul Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
no planned for now